CLINICAL TRIAL: NCT06205628
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ADX-850 in Participants With Hypertension
Brief Title: Safety, Tolerability, PK and PD of ADX-850 in Participants With Hypertension
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ADARx Pharmaceuticals, Inc. (Industry)
Collaborators: ADARx Australia Pty Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ADX-850-101
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Hypertension; Hypertension,Essential
Keywords: Hypertension
MeSH Terms: conditions — Hypertension; Essential Hypertension | interventions — RNA, Small Interfering

STUDY DESIGN:
Intervention Model Description: Model Description
Who Masked: Participant, Investigator
Masking Description: Masking Description
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADX-850 (Experimental)
  Interventions: Drug: ADX-850
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ADX-850 — siRNA duplex oligonucleotide
  Other Names: siRNA
  Arms: ADX-850
Drug: Placebo — Saline
  Arms: Placebo

SUMMARY:
This Phase 1 study will evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of ADX-850 in participants with hypertension.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) between 18 and 35 kg/m2
* Mild to moderate hypertension, mean of >130 and <165mmHg
* No use of antihypertensive medication for a minimum of 2 weeks
* Willing and able to comply with all study requirements
* Willing to take irbesartan as concomitant ARB therapy (Part 2 only)
* Must be a non-smoker for the duration of the study

Key Exclusion Criteria:

* Secondary hypertension
* Active malignancy and/or history of malignancy in the past 5 years
* History of liver disease, Gilbert's syndrome, nonalcoholic steatohepatitis, severe steatosis, or abnormal liver function test results
* Any active infection or acute illness
* Major surgery or significant traumatic injury occurring within 3 months
* Mean sitting diastolic BP (DBP) ≥110 mmHg
* Orthostatic hypotension
* Significant kidney disease or eGFR <60 mL/min/1.73m2
* Abnormal potassium levels
* History or presence of clinically significant ECG abnormalities
* Treatment with another investigational product within 30 days prior to the first study drug administration
* Pregnant, intend to become pregnant during the course of the study, or lactating
* History of alcohol abuse
* Night shift workers (regular working hours between 10:00 PM and 6:00 AM)
* Any other significant medical history, such as major cardiovascular events or cancer
* Known history of intolerance to ARB medication (Part 2 only)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-03-21 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety of ADX-850 in Participants with Hypertension | 365 days
  Incidence, relationship and severity of adverse events and serious adverse events

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of ADX-850 - Maximum Concentration | 8 days
  Cmax
Pharmacokinetics (PK) of ADX-850 - Time to Maximum Concentration | 8 days
  Tmax
Pharmacokinetics (PK) of ADX-850 - Exposure | 8 days
  Area under the Curve (AUC)
Pharmacodynamics (PD) of ADX-850 - Blood Pressure | 365 days
  Change from baseline in blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Aditya Patel, MD, Study Director — ADARx Pharmaceuticals
Locations (3):
- Australia (3):
  - CMAX Clinical Research, Adelaide, South Australia
  - Linear Clinical Research, Nedlands, Western Australia
  - Clinitrials Pty Ltd, Perth

IPD SHARING:
Plan to Share IPD: Undecided